CLINICAL TRIAL: NCT03166436
Title: Radiofrequency Ablation Plus Stenting Versus Stenting Alone for Treatment of Malignant Biliary Obstruction
Brief Title: RFA for Malignant Biliary Obstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Tomas Hucl, Vice-chairman, Department of Gastroenterology and Hepatology, Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IKEM RFA CCA PC
Record Dates: First submitted 2017-05-14; First posted 2017-05-25 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Cholangiocarcinoma; Pancreas Cancer
MeSH Terms: conditions — Cholangiocarcinoma; Pancreatic Neoplasms | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RFA plus stenting (Experimental): Endoluminal radiofrequency ablation followed by biliary stenting
  Interventions: Procedure: Radiofrequency ablation; Procedure: Biliary stenting
- Stenting alone (Active Comparator): Biliary stenting alone
  Interventions: Procedure: Biliary stenting

INTERVENTIONS:
Procedure: Radiofrequency ablation — radiofrequency ablation
  Arms: RFA plus stenting
Procedure: Biliary stenting — biliary stenting

SUMMARY:
Pancreatic cancer and cholangiocarcinoma are the most common causes of malignant biliary obstruction. They are diseases of increasing incidence and unfavorable prognosis. Only a minority of patients have a localized disease and are indicated for surgery with a chance of long-term survival. Locally advanced and metastatic tumors are treated with palliative chemotherapy or chemoradiotherapy; the results of such treatments are unsatisfactory. The average survival of patients with unresectable disease is 6 months and only 5 - 10 % of patients survive 5 years. Chemotherapy and radiotherapy can be used, however only with a palliative effect. Biliary drainage is an integral part of palliative treatment. Endoscopically or percutaneously placed stents improve quality of life, decrease cholestasis and pruritus, but do not significantly improve survival. Biliary stents get occluded over time, possibly resulting in acute cholangitis and require repeated replacement. Endoluminal biliary photodynamic therapy (PDT) and radiofrequency ablation (RFA), locally active endoscopic methods, have been increasingly used in recent years in palliative treatment of patients with malignant biliary obstruction. In photodynamic therapy, improved survival has been shown in two randomized controlled trials; however the technique suffers from technical complexity, high cost and low availability. In RFA, application of low voltage high frequency current during radiofrequency ablation results in tissue destruction by heat. Its antitumor effect may also be related to systemic changes in antitumor immunity. The use of endoluminal biliary RFA has so far been reported only in small retrospective cohorts of patients.

The aim of this randomized study is to compare efficacy of RFA plus stenting to stenting alone in palliative treatment of malignant biliary obstruction with survival as primary outcome. Secondary outcomes are stent patency, immediate and late complications, quality of life and effects on anti-tumor immunity in the RFA group.

DETAILED DESCRIPTION:
Cholangiocarcinoma and pancreatic cancer are by far the two most common causes of malignant bile duct obstruction. Cholangiocarcinoma is an adenocarcinoma originating in the bile duct whereas pancreatic cancer is an adenocarcinoma derived from pancreatic ductal cells. The incidence rates of both diseases have been rising over the past decades. Both diseases still have a very unfavorable prognosis with 5 year survival rates as low as 5-10%. Surgery represents the only therapeutic modality with a curative potential, however most patients are non-eligible for surgical treatment at the time of diagnosis. Patients present with either distant metastases, have a locally advanced disease or are unfit for surgery because of advanced age and/or co-morbidities. The prognosis of patients with unresectable bile duct or pancreatic cancer is poor with a median survival time of about 6 months. Chemotherapy and radiotherapy provide only a slight survival benefit and thus have only palliative intent.

Most patients with cholangiocarcinoma and pancreatic cancer present with bile duct obstruction in the course of their disease. Bile duct obstruction relief is an important part of palliation therapy. Endoscopic retrograde cholangiography with bile duct stenting is the method of choice with a high rate of technical success and a lower complication rate compared to surgery. Biliary stents are either plastic or metal (self-expandable metal stents, SEMS). SEMS can be covered, uncovered or partially covered. Plastic stents are cheaper and easier to exchange but have a shorter patency compared to metal stents. Metal stents have been shown to improve survival of patients with proximal malignant biliary obstruction. Both plastic and metal become occluded in a significant proportion of patients, especially in those with a longer life expectancy. Stent occlusion is often an acute event leading to sepsis and a prompt intervention is required. Failure of achieving adequate drainage may result in severe cholangitis and death.

Photodynamic therapy has been used for bile duct tumor ablation for more than a decade. It is a two stage process in which a photosensitizing agent is taken by the tumor tissue and is than activated by light of a specific wave length. Two randomized trials showed improved survival of patients treated with PDT plus stenting compared to stenting alone. However, side effects of photodynamic therapy such as phototoxicity, high costs and limited availability restrict the use of PDT.

Radiofrequency ablation (RFA), by means of alternating high-frequency current, generates heat that results in coagulation necrosis of tissue. It is widely used to treat liver tumors or dysplastic Barrett's esophagus. Endoluminal biliary RFA has become possible upon availability of narrow ERCP RFA catheters and represents a new modality of intraductal tumor ablation. The probe can be introduced over a 0.035-inch wire through a standard endoscope, thus allowing endoscopic ablation of malignant bile duct obstruction. The bipolar catheter has multiple circumferential electrodes at the distal tip. The coagulative effect is delivered in the area between the two electrodes.

A few human non-randomized case series investigating the safety and efficiency of RFA were reported. Steel at al reported their results in 22 patients with malignant bile duct obstruction (16 patients with pancreatic cancer and 6 patients with cholangiocarcinoma). Immediate, 30 day complication rates and 90 day stent patency were evaluated as primary parameters. Intraductal RFA was followed by a SEMS placement. One patient developed asymptomatic elevation of amylase, one patients developed rigors and two patients developed cholecystitis requiring cholecystectomy. All except 3 patients achieved 90 day stent patency.

In a recent study of Sharaiha et al, 26 patients with pancreatic or bile duct cancer underwent RFA followed by plastic or metal stent placement. They were compared to 40 matched controls who underwent only stenting. Technical success rate was 100%. Multivariable Cox proportional regression analysis showed RFA to be an independent predictor of survival [HR 0.29 (0.11-0.76), p = 0.012] together with age and receipt of chemotherapy [HR 1.04 (1.01-1.07), p = 0.011; HR 0.26 (0.10-0.70), p = 0.007]. Surprisingly, SEMS patency rates were the same across all groups.

In an Austrian national retrospective study, 84 ablations were performed in 58 patients in 11 centers. Cholangiocarcinoma was present in 45 patients. Technical feasibility was 100%, however multiple complications occurred (1 liver infarct, 5 cholangitis, 3 hemobilia, 2 sepsis, 1 gall-bladder empyema, 1 liver coma).

RFA was also investigated in pancreatic cancers only. In a retrospective comparison of 23 patients and 46 controls, the median survival was better in the RFA group (226 vs. 123 days, p=0,01). The median stent patency was not different.

The safety profile of RFA seems to be acceptable, however severe complications have occured. In the study of Tal et al, 3 cases of bleeding were reported, two of them resulted in death. In all of these patients, plastic stents were used.

Increasing evidence indicates that RFA might stimulate anti-tumor immunity. Active anti-cancer immune responses depend on efficient presentation of tumor antigens and cytokine-mediated stimulatory signaling. Tumor cells are generally regarded as poor stimulators of T-cells. In contrast, antigen-presenting cells (APCs) are highly specialized in this function and are therefore important in the process of stimulation of T-cell responses to tumors. RFA has been shown to stimulate anti-tumor immunity through the induction of heat shock proteins, especially HSP 70. HSPs have the capacity to affect the immunogenicity of tumor cells, to chaperone antigenic peptides and deliver them into APCs, thus activate and regulate innate and adaptive immunity.

Based on the available evidence, RFA seems to be a technically feasible technique of malignant bile duct stricture ablation with a favorable safety profile. Retrospective case series have reported improved stent patency and survival in cholangiocarcinoma and pancreatic cancer patients following RFA. Thus, endoluminal RFA may represent a novel treatment modality in patients with malignant biliary obstruction. For this to happen, however, prospectively obtained comparative data with established treatment, i.e. biliary stenting, regarding safety and efficiency are necessary.

The investigators aim to compare endoscopic radiofrequency ablation plus stenting vs. stenting alone for malignant bile duct obstruction not eligible for surgical resection in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Pathologically confirmed malignant bile duct obstruction (cholangiocarcinoma or pancreatic cancer)
* Laboratory signs of biliary obstruction
* Non-resectable disease (distant metastasis, locally advanced disease, patient related factors) based on a multidisciplinary team decision
* Capability of giving informed consent
* Life expectancy greater than 3 months

Exclusion Criteria:

* Unstable for ERC
* Inability to give informed consent
* Pregnancy
* Uncorrected coagulopathy
* Concomitant biliary oncological endoluminal therapy (photodynamic therapy, brachytherapy)
* Cardiac pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-06-08 (Estimated); Primary Completion 2019-05-08 (Estimated); Study Completion 2020-05-08 (Estimated)

PRIMARY OUTCOMES:
Survival | 12 months
  number of days/months of survival (being alive) post intervention

SECONDARY OUTCOMES:
Stent patency | 12 months
  number of days/months of patent stent (not occluded) post intervention
Complications | 30 days
  number of complications related to procedure (bleeding, perforation, cholangitis will be combined to report as a complication)
Quality of life | 12 months
  validated questionnaire investigating quality of live post intervention
Augmentation of antitumor immunity | 30 days
  serum level of HSP 70 and selected cytokines will be measured from blood

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Hucl, MD, PhD, Principal Investigator — Institute for Clinical and Experimental Medicine
Locations (1):
- Department of Gastroenterology and Hepatology, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ilyas SI, Gores GJ. Pathogenesis, diagnosis, and management of cholangiocarcinoma. Gastroenterology. 2013 Dec;145(6):1215-29. doi: 10.1053/j.gastro.2013.10.013. Epub 2013 Oct 15. PMID 24140396
- [Background] Khan SA, Davidson BR, Goldin RD, Heaton N, Karani J, Pereira SP, Rosenberg WM, Tait P, Taylor-Robinson SD, Thillainayagam AV, Thomas HC, Wasan H; British Society of Gastroenterology. Guidelines for the diagnosis and treatment of cholangiocarcinoma: an update. Gut. 2012 Dec;61(12):1657-69. doi: 10.1136/gutjnl-2011-301748. Epub 2012 Aug 15. PMID 22895392
- [Background] Rerknimitr R, Angsuwatcharakon P, Ratanachu-ek T, Khor CJ, Ponnudurai R, Moon JH, Seo DW, Pantongrag-Brown L, Sangchan A, Pisespongsa P, Akaraviputh T, Reddy ND, Maydeo A, Itoi T, Pausawasdi N, Punamiya S, Attasaranya S, Devereaux B, Ramchandani M, Goh KL; Asia-Pacific Working Group on Hepatobiliary Cancers. Asia-Pacific consensus recommendations for endoscopic and interventional management of hilar cholangiocarcinoma. J Gastroenterol Hepatol. 2013 Apr;28(4):593-607. doi: 10.1111/jgh.12128. PMID 23350673
- [Background] Vincent A, Herman J, Schulick R, Hruban RH, Goggins M. Pancreatic cancer. Lancet. 2011 Aug 13;378(9791):607-20. doi: 10.1016/S0140-6736(10)62307-0. Epub 2011 May 26. PMID 21620466
- [Background] Davids PH, Groen AK, Rauws EA, Tytgat GN, Huibregtse K. Randomised trial of self-expanding metal stents versus polyethylene stents for distal malignant biliary obstruction. Lancet. 1992 Dec 19-26;340(8834-8835):1488-92. doi: 10.1016/0140-6736(92)92752-2. PMID 1281903
- [Background] Sangchan A, Kongkasame W, Pugkhem A, Jenwitheesuk K, Mairiang P. Efficacy of metal and plastic stents in unresectable complex hilar cholangiocarcinoma: a randomized controlled trial. Gastrointest Endosc. 2012 Jul;76(1):93-9. doi: 10.1016/j.gie.2012.02.048. Epub 2012 May 15. PMID 22595446
- [Background] Ortner ME, Caca K, Berr F, Liebetruth J, Mansmann U, Huster D, Voderholzer W, Schachschal G, Mossner J, Lochs H. Successful photodynamic therapy for nonresectable cholangiocarcinoma: a randomized prospective study. Gastroenterology. 2003 Nov;125(5):1355-63. doi: 10.1016/j.gastro.2003.07.015. PMID 14598251
- [Background] Zoepf T, Jakobs R, Arnold JC, Apel D, Riemann JF. Palliation of nonresectable bile duct cancer: improved survival after photodynamic therapy. Am J Gastroenterol. 2005 Nov;100(11):2426-30. doi: 10.1111/j.1572-0241.2005.00318.x. PMID 16279895
- [Background] Curley SA, Izzo F. Radiofrequency ablation of primary and metastatic hepatic malignancies. Int J Clin Oncol. 2002 Apr;7(2):72-81. doi: 10.1007/s101470200010. PMID 12018113
- [Background] Shaheen NJ, Overholt BF, Sampliner RE, Wolfsen HC, Wang KK, Fleischer DE, Sharma VK, Eisen GM, Fennerty MB, Hunter JG, Bronner MP, Goldblum JR, Bennett AE, Mashimo H, Rothstein RI, Gordon SR, Edmundowicz SA, Madanick RD, Peery AF, Muthusamy VR, Chang KJ, Kimmey MB, Spechler SJ, Siddiqui AA, Souza RF, Infantolino A, Dumot JA, Falk GW, Galanko JA, Jobe BA, Hawes RH, Hoffman BJ, Sharma P, Chak A, Lightdale CJ. Durability of radiofrequency ablation in Barrett's esophagus with dysplasia. Gastroenterology. 2011 Aug;141(2):460-8. doi: 10.1053/j.gastro.2011.04.061. Epub 2011 May 6. PMID 21679712
- [Background] Zacharoulis D, Lazoura O, Sioka E, Potamianos S, Tzovaras G, Nicholls J, Koukoulis G, Habib N. Habib EndoHPB: a novel endobiliary radiofrequency ablation device. An experimental study. J Invest Surg. 2013 Feb;26(1):6-10. doi: 10.3109/08941939.2012.681832. Epub 2012 Dec 28. PMID 23273142
- [Background] Steel AW, Postgate AJ, Khorsandi S, Nicholls J, Jiao L, Vlavianos P, Habib N, Westaby D. Endoscopically applied radiofrequency ablation appears to be safe in the treatment of malignant biliary obstruction. Gastrointest Endosc. 2011 Jan;73(1):149-53. doi: 10.1016/j.gie.2010.09.031. PMID 21184881
- [Background] Sharaiha RZ, Natov N, Glockenberg KS, Widmer J, Gaidhane M, Kahaleh M. Comparison of metal stenting with radiofrequency ablation versus stenting alone for treating malignant biliary strictures: is there an added benefit? Dig Dis Sci. 2014 Dec;59(12):3099-102. doi: 10.1007/s10620-014-3264-6. Epub 2014 Jul 18. PMID 25033929
- [Background] Monga A, Gupta R, Ramchandani M, Rao GV, Santosh D, Reddy DN. Endoscopic radiofrequency ablation of cholangiocarcinoma: new palliative treatment modality (with videos). Gastrointest Endosc. 2011 Oct;74(4):935-7. doi: 10.1016/j.gie.2010.10.018. Epub 2010 Dec 18. No abstract available. PMID 21168839
- [Background] Dolak W, Schreiber F, Schwaighofer H, Gschwantler M, Plieschnegger W, Ziachehabi A, Mayer A, Kramer L, Kopecky A, Schrutka-Kolbl C, Wolkersdorfer G, Madl C, Berr F, Trauner M, Puspok A; Austrian Biliary RFA Study Group. Endoscopic radiofrequency ablation for malignant biliary obstruction: a nationwide retrospective study of 84 consecutive applications. Surg Endosc. 2014 Mar;28(3):854-60. doi: 10.1007/s00464-013-3232-9. Epub 2013 Oct 3. PMID 24196547
- [Background] Kallis Y, Phillips N, Steel A, Kaltsidis H, Vlavianos P, Habib N, Westaby D. Analysis of Endoscopic Radiofrequency Ablation of Biliary Malignant Strictures in Pancreatic Cancer Suggests Potential Survival Benefit. Dig Dis Sci. 2015 Nov;60(11):3449-55. doi: 10.1007/s10620-015-3731-8. Epub 2015 Jun 3. PMID 26038094
- [Background] Tal AO, Vermehren J, Friedrich-Rust M, Bojunga J, Sarrazin C, Zeuzem S, Trojan J, Albert JG. Intraductal endoscopic radiofrequency ablation for the treatment of hilar non-resectable malignant bile duct obstruction. World J Gastrointest Endosc. 2014 Jan 16;6(1):13-9. doi: 10.4253/wjge.v6.i1.13. PMID 24527176
- [Background] Wu F. Heat-Based Tumor Ablation: Role of the Immune Response. Adv Exp Med Biol. 2016;880:131-53. doi: 10.1007/978-3-319-22536-4_8. PMID 26486336
- [Background] Witzigmann H, Berr F, Ringel U, Caca K, Uhlmann D, Schoppmeyer K, Tannapfel A, Wittekind C, Mossner J, Hauss J, Wiedmann M. Surgical and palliative management and outcome in 184 patients with hilar cholangiocarcinoma: palliative photodynamic therapy plus stenting is comparable to r1/r2 resection. Ann Surg. 2006 Aug;244(2):230-9. doi: 10.1097/01.sla.0000217639.10331.47. PMID 16858185
- [Derived] Jarosova J, Zarivnijova L, Cibulkova I, Mares J, Macinga P, Hujova A, Falt P, Urban O, Hajer J, Spicak J, Hucl T. Endoluminal radiofrequency ablation in patients with malignant biliary obstruction: a randomised trial. Gut. 2023 Nov 24;72(12):2286-2293. doi: 10.1136/gutjnl-2023-329700. PMID 37652677